CLINICAL TRIAL: NCT01119586
Title: Identifying Rare Genetic Variants Involved in High Risk Acute Lymphoblastic Leukemia (ALL) Via Pooled DNA Sequencing
Brief Title: Biomarkers in DNA Samples From Patients With High-Risk Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL10B2; COG-AALL10B2 (Other: Children's Oncology Group); CDR0000672526 (Other: Clinicaltrials.gov); NCI-2011-02232 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: B-cell adult acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Genetic Linkage; Microarray Analysis; Base Sequence; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: genetic linkage analysis
Genetic: microarray analysis
Genetic: nucleic acid sequencing
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood or tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in DNA samples from patients with newly diagnosed high-risk acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To perform pooled DNA sequencing in 56 genes from the genomic DNA of unaffected children and matched non-tumor and blast DNA from patients with high-risk (HR) acute lymphoblastic leukemia (ALL) enrolled on COG HR ALL protocols.
* To identify loci enriched for genetic variation between DNA of unaffected children and DNA of these patients.
* To individually validate novel, putatively functional single nucleotide polymorphisms (SNPs) identified via pooled sequencing with another genotyping platform.
* To correlate HR ALL with clinical phenotypes, co-morbidities, toxicities, outcomes to the genes or pathways found to harbor a significant increase in genetic variation.

OUTLINE: DNA specimens from unaffected children (pool 1) and from patients with non-tumor (pool 2) and leukemia blasts (pool 3) are analyzed for genetic pathophysiology of pre-B acute lymphoblastic leukemia by microarray and PCR assays. Sequencing is performed on each of the 3 PCR pools of DNA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed with high-risk B-precursor acute lymphoblastic leukemia

  * Matched patients non-tumor and blast DNA samples
  * Enrolled on COG-P9906 or COG-AALL0232 protocols
* Cohort of random pediatric DNA samples extracted from newborn infants' blood spots from the State of Missouri

PATIENT CHARACTERISTICS:

* Newborn infants from the state of Missouri

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients With High-Risk Acute Lymphoblastic Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Identification of loci enriched for genetic variation suggestive of pre-B leukemogenesis
Correlation between high-risk acute lymphoblastic leukemia with clinical phenotypes, co-morbidities, toxicities, outcomes to the genes or pathways found to harbor a significant increase in genetic variation

CONTACTS AND LOCATIONS:
Overall Officials: Todd E. Druley, MD, Principal Investigator — St. Louis Children's Hospital